CLINICAL TRIAL: NCT04374344
Title: Qualitative Analysis of Photoplethysmography Waveforms for the Detection of Cardiac Arrhythmias Using a Pulse-deriving Smartphone Application
Brief Title: Qualitative Analysis of Photoplethysmography Waveforms for the Detection of Cardiac Arrhythmias
Acronym: INTERPRET-AF I
Status: Completed | Type: Observational
Sponsor: Qompium NV (Industry)
Responsible Party: Sponsor
Other Study IDs: 3
Record Dates: First submitted 2020-04-28; First posted 2020-05-05 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Cardiac Arrhythmia
Keywords: Qualitative analysis; Photoplethysmography; Single-lead electrocardiography
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical professionals: Medical professionals including cardiologists and cardiology residents.
  Interventions: Other: Qualitative analysis of PPG, single-lead ECG, and 12-lead ECG measurements

INTERVENTIONS:
Other: Qualitative analysis of PPG, single-lead ECG, and 12-lead ECG measurements — Participants are instructed to qualitatively analyse PPG, single-lead ECG, and 12-lead ECG heart rhythm traces.

SUMMARY:
Single-lead electrocardiography (ECG) technologies and photoplethysmography (PPG) deriving smartphone apps are gaining interest in the heart rhythm detection space since these apps have the potential to capture and assess heart rhythms. Proprietary arrhythmia detection algorithms are proven to be reliable and accurate. However, insights into the readability of PPG waveforms by human reviewers remain limited. To the investigators' knowledge, there are no publications available regarding the readability of PPG waveforms by human reviewers. The objective of the study was to assess the readability of PPG and single-lead ECG analysis by medical professionals, with respect to the gold-standard 12-lead ECG diagnosis, and investigate whether additional information positively impacts PPG analysis.

DETAILED DESCRIPTION:
During the study, the readability of PPG and single-lead ECG waveform analysis will be investigated. The objective of the study is to determine the readability of PPG and single-lead ECG measurements, with respect to the gold-standard 12-lead ECG, and investigate whether additional information positively impacts the readability of PPG. Medical professionals (cardiologists and cardiology residents), blinded for the patients' characteristics and history, are instructed to separately analyse the following signals, obtained from 30 patients.

* 30 outputs with PPG waveforms
* 30 outputs with PPG waveforms with tachogram and Poincaré
* 30 outputs with PPG waveforms with tachogram, Poincaré, and algorithm interpretation
* 30 outputs with single-lead ECG waveforms
* 30 outputs with 12-lead ECG waveforms

Participants report the results of the qualitative analysis via a digital questionnaire with multiple-choice questions. Medical professionals classify each rhythm trace as regular rhythm, one or more ectopic/missed heartbeats, atrial flutter, atrial fibrillation, unreadable, or other. The tachogram, Poincaré, and the algorithm interpretation are subsequently added to investigate whether the additional information improves the readability of PPG. Based on the provided answers, the study team will determine the readability of PPG and single-lead ECG analysis interpretation, with respect to the gold-standard 12-lead ECG diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Cardiologist or cardiology resident
* Able to understand Dutch or English

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Medical professionals including cardiologists and cardiology residents with and without experience in qualitative analysis of PPG waveforms.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy to discriminate between atrial fibrillation and non-atrial fibrillation rhythms | Through study completion, an average of 3 months
  Readability assessment (sensitivity, specificity, positive predictive value, negative predictive value, and accuracy) of PPG and single-lead ECG signals to detect atrial fibrillation. The readability will be determined and compared with the gold-standard 12-lead ECG diagnosis.

SECONDARY OUTCOMES:
Required elements to increase the readability of PPG measurements | Through study completion, an average of 3 months
  Readability assessment (sensitivity, specificity, positive predictive value, negative predictive value, and accuracy) of PPG waveforms, PPG waveforms with tachogram and Poincaré, and PPG waveforms with tachogram, Poincaré and algorithm interpretation. The readability will be determined and compared with the gold-standard 12-lead ECG diagnosis.
Diagnostic accuracy of PPG analysis: experienced in PPG analysis vs inexperienced in PPG analysis | Through study completion, an average of 3 months
  Readability assessment (sensitivity, specificity, positive predictive value, negative predictive value, and accuracy) of PPG waveforms, PPG waveforms with tachogram and Poincaré, and PPG waveforms with tachogram, Poincaré and algorithm interpretation. The readability will be determined and compared with the gold-standard 12-lead ECG diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Vandervoort, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided